CLINICAL TRIAL: NCT05226221
Title: Mortality and Morbidity in Emergency Gastrointestinal Surgery: Comparison of Different Incidence of Interventions According to the ICD-9-CM Classification in Relation to the Age Groups
Brief Title: Gastrointestinal Emergency Surgery: Evaluation of Morbidity and Mortality
Acronym: GESEMM
Status: Recruiting | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Gianluca Costa, MD, PhD, Campus Bio-Medico University
Other Study IDs: 87/21 (OSS)
Record Dates: First submitted 2022-01-18; First posted 2022-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Injury; Gastrointestinal Hemorrhage; Gastrointestinal Lesions; Gastrointestinal Ulcer; Gastrointestinal Perforation; Gastrointestinal Cancer
Keywords: gastrointestinal emergency, acute care surgery
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal Emergency Surgery: Evaluation of Morbidity and Mortality

DETAILED DESCRIPTION:
Background: Gastrointestinal emergencies (GE) are frequently encountered in the emergency department (ED), and patients can present with wide-ranging symptoms. Symptoms that suggest an underlying GE can include: abdominal pain; nausea; vomiting; diarrhoea; melaena; haematemesis; constipation; jaundice; and abdominal distension. Abdominal pain is a common ED presentation and can be the cause of a wide variety of GE. The acute abdomen (AB) is a term given to sudden severe pain in the abdomen requiring fast diagnosis and treatment usually requiring emergency surgical procedures. Causes of AB may include: appendicitis; pancreatitis; peptic ulcer disease (PUD); gall bladder pathology; intestinal ischemia; diverticulitis; intestinal obstruction; and ruptured ectopic pregnancy. Emergency gastrointestinal surgery (EGS) is burdened by significant mortality and morbidity rates because it is performed with little to no advance planning or preparation, on patients who are in dire straits. Scott JW et al report that there are more than 3 million patients admitted to US hospitals each year for EGS diagnoses, more than the sum of all new cancer diagnoses. (Scotte JW) In addition to the complexity of the urgent surgical patient (often suffering from multiple co-morbidities), there is the unpredictability and the severity of the event. Frequently, it is necessary rapid decision-making that allows a correct diagnosis and an adequate and timely treatment. (See Ref.) Moreover, another study by Havens JM et al reported that patients undergoing EGS operation are up to 8 times more likely to die postoperatively than are patients undergoing the same procedures electively. Furthermore, the increase in average life will lead more and more people over 65 to face surgical pathologies in an emergency setting, and in the elderly EGS is characterized by greater morbidity and mortality as well as by a global worsening of the residual quality of life (QoL). The explanation for the high percentage of acute complications could be found in the inevitable reduction of the functional reserve related to age. An example is the reduction of the body's immune defenses in the humoral response of B cells, in the cell-mediated immune function and macrophage activity which explains the susceptibility to infectious complications, facilitated by the altered integrity of the skin barrier and mucous membranes too. Is in this setting that tools capable to help the surgeon in the decision-making process in order to reduce mortality and morbidity linked to the EGS could become very useful. To do this, it is necessary to study the greatest number of risk factors associated with EGS, considering all age groups and all types of diseases.

AIM: To analyze the clinicopathological findings, management strategies, and short-term outcomes of gastrointestinal emergency procedures; to evaluate the prognostic role of existing risk-scores; to define the most suitable scoring system or gastro-intestinal surgical emergency; to identify any specific parameters that may be used as variables for a new scoring system, peri-operative variables predicting adverse results and any critical issues in the management of these patients.

STUDY DESIGN: both retrospective and prospective cohort, multicenter, observational, no profit clinical study. All the study participants will collect data on > 18 y. o. patients underwent general emergency surgery during an 18 month period, guaranteeing whole completeness of the picked data > 95%. This study was approved by the Health Sciences Research Ethics Board of the University Campus Biomedio of Rome

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. completed at the day of surgery
* Emergency gastrointestinal surgery considered as not-scheduled procedure

Exclusion Criteria:

* Age under 18 y.o. at the day of surgery
* Lack of informed consent
* Patients already hospitalized and scheduled for the same procedure
* Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter italian national survey cohort study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality rate | 18 months
  any cause of mortality related to surgical procedure
30-day morbidity rate | 18 months
  Morbidity defined by mean of the Clavien's Classification scoring system

SECONDARY OUTCOMES:
Calculation of Charlson Age-Comorbidity Index (CACI) | 8 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Simplified Acute Physiology Score-II (SAPS-II) | 18 months
  Calculation and evaluation of its predictive value for mortality
American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) surgical risk calculator | 18 months
  Calculation and evaluation of its predictive value for post-operative complications
5-item Frailty Index | 18 months
  Frailty stratification in participants
Total number of subjects underwent emergency surgery | 18 months
  Number of patients submitted to surgery
Emergency Surgical Frailty Index (EmFSI) | 18 months
  Frailty stratification in participants

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Biomedico, Rome, Lazio, Italy

REFERENCES:
- [Result] Fransvea P, Fico V, Cozza V, Costa G, Lepre L, Mercantini P, La Greca A, Sganga G; ERASO study group. Clinical-pathological features and treatment of acute appendicitis in the very elderly: an interim analysis of the FRAILESEL Italian multicentre prospective study. Eur J Trauma Emerg Surg. 2022 Apr;48(2):1177-1188. doi: 10.1007/s00068-021-01645-9. Epub 2021 Mar 18. PMID 33738537
- [Result] Costa G, Bersigotti L, Massa G, Lepre L, Fransvea P, Lucarini A, Mercantini P, Balducci G, Sganga G, Crucitti A; ERASO (Elderly Risk Assessment, Surgical Outcome) Collaborative Study Group. The Emergency Surgery Frailty Index (EmSFI): development and internal validation of a novel simple bedside risk score for elderly patients undergoing emergency surgery. Aging Clin Exp Res. 2021 Aug;33(8):2191-2201. doi: 10.1007/s40520-020-01735-5. Epub 2020 Nov 18. PMID 33205380
- [Result] Ceresoli M, Carissimi F, Nigro A, Fransvea P, Lepre L, Braga M, Costa G; List of Elderly Risk Assessment and Surgical Outcome (ERASO) Collaborative Study Group endorsed by SICUT, ACOI, SICG, SICE, and Italian Chapter of WSES. Emergency hernia repair in the elderly: multivariate analysis of morbidity and mortality from an Italian registry. Hernia. 2022 Feb;26(1):165-175. doi: 10.1007/s10029-020-02269-5. Epub 2020 Jul 31. PMID 32737706
- [Result] Fransvea P, Costa G, Lepre L, Podda M, Giordano A, Bellanova G, Agresta F, Marini P, Sganga G; ERASO (Elderly Risk Assessment and Surgical Outcome) Collaborative Study Group. Laparoscopic Repair of Perforated Peptic Ulcer in the Elderly: An Interim Analysis of the FRAILESEL Italian Multicenter Prospective Cohort Study. Surg Laparosc Endosc Percutan Tech. 2020 Jul 14;31(1):2-7. doi: 10.1097/SLE.0000000000000826. PMID 32675754
- [Result] Costa G, Fransvea P, Podda M, Pisanu A, Carrano FM, Iossa A, Balducci G, Agresta F; ERASO (Elderly Risk Assessment and Surgical Outcome) Collaborative Study Group. The use of emergency laparoscopy for acute abdomen in the elderly: the FRAILESEL Italian Multicenter Prospective Cohort Study. Updates Surg. 2020 Jun;72(2):513-525. doi: 10.1007/s13304-020-00726-5. Epub 2020 Feb 22. PMID 32088854